CLINICAL TRIAL: NCT05367180
Title: Impact of a Prevention Program on Sun Risks in Primary School in Tropical French Region
Brief Title: The Impact of a Prevention Program on Sun Risks in Primary School in Tropical French Region
Acronym: PRESOLRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022/CHU/09
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-10

CONDITIONS: Melanoma
Keywords: School; Environment; Preventive medicine and public health; Children's health; Sun protection factor
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reference Arm (No Intervention): no preventive action
- Vivre avec le Soleil (Experimental): Use of existing validated program "vivre avec le soleil"
  Interventions: Other: "Vivre avec le Soleil" prevention program on sun risks
- Vivre avec le Soleil + program of MISOLRE association (Experimental): Use of existing validated program "vivre avec le soleil" associated with prevention awareness program of MISOLRE association
  Interventions: Other: MISOLRE prevention program on sun risks; Other: "Vivre avec le Soleil" prevention program on sun risks
- Vivre avec le Soleil + program of MISOLRE association + sun protections (Experimental): Use of existing validated program "vivre avec le soleil" associated with prevention awareness program of MISOLRE association and with the distribution of caps, sunscreens and sunglasses
  Interventions: Other: MISOLRE prevention program on sun risks; Other: "Vivre avec le Soleil" prevention program on sun risks; Other: Sun protection equipment

INTERVENTIONS:
Other: MISOLRE prevention program on sun risks — Training of an ambassador class by a field coordinator Dissemination of the information by the ambassador class to the other classes of the school drawn by lot Transmission of an information document to parents on photoprotection to make them aware of the actions to adopt
  Arms: Vivre avec le Soleil + program of MISOLRE association; Vivre avec le Soleil + program of MISOLRE association + sun protections
Other: "Vivre avec le Soleil" prevention program on sun risks — Program is delivered directly by the teachers through pedagogical books : 10 workshops over a period of 3 months
  Arms: Vivre avec le Soleil; Vivre avec le Soleil + program of MISOLRE association; Vivre avec le Soleil + program of MISOLRE association + sun protections
Other: Sun protection equipment — Distribution of sunscreen, caps and sunglasses
  Arms: Vivre avec le Soleil + program of MISOLRE association + sun protections

SUMMARY:
Sun exposure during childhood can cause the development of skin cancer in later years, in particular melanoma, which is the most lethal.The worldwide incidence of melanoma is on the rise, with nearly 290,000 new cases diagnosed in 2018. The country with the highest age-standardized incidence rate is Australia, where 40.4 cases per 100,000 men and 27.5 cases per 100,000 women were reported in 2018. Since 2008, however, this incidence has decreased by 11% in the 14-49 age group following the implementation of effective sun safety campaigns. In the French overseas department of Reunion Island, which is characterized by a great diversity of skin phototypes due to multiple migratory flows, the ultraviolet (UV) index is very high - equivalent to that in Australia. The age-standardized incidence rate of melanoma Reunion Island increased fourfold between 1995 and 2015. In 2015, it was estimated at nearly 30.0 new cases per 100,000 inhabitants in people with skin phototypes I-III, compared to 13.5 in metropolitan France.

Over the course of a lifetime, 80% of exposure to UV radiation and 50% of skin damage occur before the age of 21, mainly in the school environment. In spite of this, knowledge of the risks associated with sun exposure remains insufficient among children and adolescents. Similar quantitative data have been reported for Reunion Island by the local association MiSolRé (Mission Soleil Réunion), which has been running sun safety campaigns in elementary schools since 2017. However, methodological limitations compromise the validity and extrapolation of the results. And the question arises as to the type of programme to be implemented: strengthening individual skills through health education methods? Community reinforcement through training activities involving peers? Improving access to prevention? Thus, it seems necessary to rigorously evaluate the effectiveness of different actions such as the educational programme "Vivre avec le soleil" alone or associated with the visit of professionals in the field with or without distribution of photoprotection material. The aim of this randomized controlled trial is to evaluate the effectiveness of three awareness-raising programmes on the risks linked to sun exposure, delivered in primary school classes in Reunion Island, on the pupils' knowledge of sun prevention.

ELIGIBILITY:
Inclusion Criteria:

* students in a primary school in Reunion Island, drawn by lot for the study and whose school director agrees to participate in the program
* in a primary school with more than 10 classes
* within a class from the second and the third cycle: CE (elementary course) 1, CE2, CM (average course) 1 or CM2
* whose 2 parents have given their consent

Exclusion Criteria:

* in a school that has already benefited from the awareness program by the MiSolRé association in 2016/2017, 2017/2018, 2019/2020, 2020/2021
* in CP (preparatory course) class
* in a multi-level class

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1452 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of 3 programs of awareness of the risks related to sun exposure, delivered in primary school classes in Reunion Island, on students' knowledge of sun prevention | 6 months after inclusion
  self questionnaire completed by the students. Comparison of pourcentage of good response to knowledge questionnaire in the 4 arms. No minimum or maximum score.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BERTOLOTTI, Principal Investigator — CHU de La Réunion
Locations (1):
- CHU de La Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dugast C, Bruneau L, Fianu A, Ferdynus C, Boussaid K, Vuichard J, Duloutre F, Dumez J, Sultan-Bichat N, Bertolotti A. PRESOLRE: study protocol for a primary school-based, cluster randomised controlled trial of three sun exposure risk prevention strategies on Reunion Island. BMJ Open. 2024 May 15;14(5):e082045. doi: 10.1136/bmjopen-2023-082045. PMID 38754877